CLINICAL TRIAL: NCT01574651
Title: A 26-week Treatment, Multicenter, Randomized, Parallel Group, Blinded Study to Assess the Efficacy and Safety of QVA149 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease Using Tiotropium Plus Formoterol as Control
Brief Title: The Effect of QVA149 on Health Related Quality of Life in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: QUANTIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149ADE01; 2011-004870-26 (EudraCT Number)
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: QVA149; Health related quality of life; Formoterol; Tiotropium; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 plus placebo to tiotropium and placebo to formoterol (Experimental): QVA149 110/50µg, once daily for inhalation use plus placebo to tiotropium, once daily for inhalation use and placebo to formoterol, twice daily for inhalation use.
  Interventions: Drug: QVA149; Drug: Placebo to tiotropium; Drug: Placebo to formoterol
- Tiotropium plus Formoterol and placebo to QVA149 (Active Comparator): Tiotropium 18µg, once daily for inhalation use plus Formoterol 12µg, twice daily for inhalation use and placebo to QVA149, once daily for inhalation use.
  Interventions: Drug: Tiotropium; Drug: Formoterol; Drug: Placebo to QVA149

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50µg, once daily (q.d.) is administered via a single-dose dry powder inhaler
  Arms: QVA149 plus placebo to tiotropium and placebo to formoterol
Drug: Placebo to tiotropium — Placebo to tiotropium capsules daily (q.d.) for inhalation, delivered via proprietary inhaler (Handihaler®). Placebo tiotropium inhalation capsules were matched in size and color to tiotropium 18 μg q.d. inhalation capsules
  Arms: QVA149 plus placebo to tiotropium and placebo to formoterol
Drug: Placebo to formoterol — Placebo to formoterol capsules twice daily (b.i.d) delivered via Aerolizer® device. Placebo formoterol inhalation capsules were equally matched in size, shape and color to formoterol 12 μg b.i.d. inhalation capsules.
  Arms: QVA149 plus placebo to tiotropium and placebo to formoterol
Drug: Tiotropium — Tiotropium 18µg, once daily is administered via the manufacturer's proprietary inhalation device.
  Arms: Tiotropium plus Formoterol and placebo to QVA149
Drug: Formoterol — Formoterol 12µg, twice daily is administered via the manufacturer's proprietary inhalation device.
  Arms: Tiotropium plus Formoterol and placebo to QVA149
Drug: Placebo to QVA149 — Placebo to QVA149 is administered via a single-dose dry powder inhaler. Placebo QVA149 inhalation capsules were equally matched in size, shape and color to QVA149 110/50 μg q.d. inhalation capsules
  Arms: Tiotropium plus Formoterol and placebo to QVA149

SUMMARY:
This study will assess the efficacy and safety of QVA149 compared to tiotropium plus formoterol in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 40 yrs
* Patients with moderate to severe chronic obstructive pulmonary disease (GOLD 2010 guidelines)
* Smoking history of at least 10 pack years
* Post-bronchodilator FEV1 < 80% and ≥30% of the predicted normal value and post-bronchodilator FEV1/FVC (forced vital capacity) <70%

Exclusion Criteria:

* Pregnant women or nursing mothers or women of child-bearing potential not using adequate contraception
* Patients with a history of long QT syndrome
* Patients with Type I or uncontrolled Type II diabetes
* Patients who have had a COPD exacerbation or respiratory tract infection within 6 weeks prior to screening
* Patients with any history of asthma
* Patients with pulmonary lobectomy, lung volume reduction surgery, or lung transplantation
* Patients with concomitant pulmonary disease
* Patients requiring long term oxygen therapy (>15 h a day)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (113):
- Germany (113):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Heidelberg, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Teterow, Germany
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Neustadt an der Saale
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Bergisch Gladbach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borna
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Donaustauf
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eggenfelden
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Eschwege
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Euskirchen
  - Novartis Investigative Site, Forchheim
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Geesthacht
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Güstrow
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hannover Münden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hettstedt
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Höchstadt an der Aisch
  - Novartis Investigative Site, Kamen
  - Novartis Investigative Site, Kamenz
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Menden
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Oranienburg
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Oschersleben
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Peine
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien A. Chiemsee
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Rathenow
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Roth
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Schwabach
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Sonneberg
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Teuchern
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Vöhringen
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Weyhe
  - Novartis Investigative Site, Wiesloch
  - Novartis Investigative Site, Wissen
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Zerbst

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Started | 476 | 458
Full Analysis Set (FAS) | 476 | 458
Per Protocol Set (PPS) | 373 | 374
Completed | 415 | 406
Not Completed | 61 | 52
Not completed — Lost to Follow-up | 2 | 4
Not completed — Administrative problems | 0 | 1
Not completed — Death | 3 | 3
Not completed — Patient's inability to use the device | 0 | 1
Not completed — Adverse Event | 36 | 27
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Abnormal test procedure result(s) | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 6 | 0
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149 | Total
Number analyzed (Participants) | 476 | 458 | 934
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (8.43) | 63.1 (8.15) | 62.9 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 160 | 319
  Male | 317 | 298 | 615

OUTCOME MEASURES:

1. Primary Outcome: St. George's Respiratory Questionnaire (SGRQ-C) Total Score After 26 Weeks of Treatment (Non-inferiority Analysis).
Description: SGRQ is a health related quality of life questionnaire consisting of 40 items in three areas: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). The total score is 0 to 100 with a higher score indicating poorer health status. For patients who completed the study but with missing SGRQ-C during treatment, the missing SGRQ-C were replaced by the last observation carried forward (LOCF). Symptom scores were expected to improve over treatment, therefore the replacement of missing values with earlier measurements did not result in overoptimistic imputation and this procedure could be regarded as conservative.
Time Frame: Baseline, week 26
Population: Full analysis set (FAS): all randomized patients who received at least one dose of randomized study drug. Following the ITT principle, patients were analyzed according to the treatment they were assigned to. The FAS was used for all efficacy variables unless otherwise stated.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Score on a scale
  Baseline (n=452,441) | 44.70 (17.718) | 45.68 (17.720)
  Week 26 (n=475,456) | 41.30 (19.923) | 43.19 (19.284)

2. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ-C) Total Score After 26 Weeks of Treatment (Superiority Analysis).
Description: SGRQ is a health related quality of life questionnaire consisting of 40 items in three areas: symptoms (respiratory symptoms and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). The total score is 0 to 100 with a higher score indicating poorer health status. For patients who completed the study but with missing SGRQ-C during treatment, the missing SGRQ-C were replaced by the last observation carried forward (LOCF). Symptom scores were expected to improve over treatment, therefore the replacement of missing values with earlier measurements did not result in overoptimistic imputation and this procedure could be regarded as conservative. Superiority of QVA 110/50 μg to tiotropium 18 μg q.d. plus formoterol 12 μg b.i.d. in terms of health related quality of life as assessed by St George's Respiratory Questionnaire (SGRQ-C) after 26 weeks of treatment
Time Frame: Baseline, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Score on a scale
  Baseline (n=452,441) | 44.70 (17.718) | 45.68 (17.720)
  Week 26 (n=475,456) | 41.30 (19.923) | 43.19 (19.284)

3. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score After 26 Weeks of Treatment.
Description: Baseline Dyspnea Index (BDI)/Transition Dyspnea Index (TDI) focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. BDI was measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best). TDI captures changes from baseline. Each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score. missing values were replaced by the latest observed value (LOCF)
Time Frame: Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 462 | 443
Units on a scale | 1.34 (3.440) | 0.87 (3.439)

4. Secondary Outcome: Percent of Participants With at Least One Exacerbation Requiring Systemic Corticosteroids and/or Antibiotics Over 26 Weeks
Description: The percent of participants with at least one moderate exacerbation within the 26 weeks that required systemic corticosteroids and/or antibiotics during the treatment
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Percent of participants | 10.9 | 13.3

5. Secondary Outcome: Percent of Participants With at Least One Exacerbation Requiring Hospitalization
Description: The percent of patients with at least one severe exacerbation within the 26 weeks that required hospitalization. COPD exacerbations were considered to be severe if hospitalization were required.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Percent of participants | 2.1 | 2.4

6. Secondary Outcome: Time- Event Analysis, Number of Participants With at Least One COPD Exacerbation (Moderate or Severe) During the Treatment Period
Description: The number of participants with at least one moderate or severe COPD exacerbation. COPD exacerbations are considered to be moderate if treatment with systemic corticosteroids and/or antibiotics was required. COPD exacerbations are considered to be severe if hospitalizations were required.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Participants | 62 | 70

7. Secondary Outcome: Trough FEV1 at Baseline and Week 26
Description: Trough FEV1 is the mean value of FEV1 (forced expiratory volume in one second) measured at 23:15h and 23:45h after the morning doses. The baseline value was measured at day 1 prior to the first dose.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Liters
  Baseline | 1.329 (0.4806) | 1.313 (0.4525)
  Week 26 | 1.495 (0.5060) | 1.409 (0.4878)

8. Secondary Outcome: FEV1 30 Min After the Morning Dose at Baseline and Week 26
Description: FEV1 30min is the forced expiratory volume in one second measured 30 min after the morning dose.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Liters
  Baseline (n=475,458) | 1.517 (0.5025) | 1.495 (0.4860)
  Week 26 (n=476,458) | 1.605 (0.5356) | 1.565 (0.5124)

9. Secondary Outcome: Symptoms Score Reported by the Patients Using Part I "Symptoms" of SGRO-C
Description: Part I of the SGRQ-C covers "symptoms" and is concerned with respiratory symptoms, their frequency and severity. Each questionnaire response has a unique empirically derived "weight". A score was calculated from these weights. The lowest possible value is zero and the highest 100. A higher value corresponds to greater impairment of health status.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Number analyzed (Participants) | 476 | 458
Score on a scale
  Baseline (n=473,457) | 64.10 (19.884) | 64.29 (19.768)
  Week 26 (n=476,458) | 58.31 (21.764) | 60.16 (20.678)

ADVERSE EVENTS:
Arm/Group | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol | Tiotropium Plus Formoterol and Placebo to QVA149
Serious Adverse Events (participants affected / at risk) | 30/476 | 24/458
Other Adverse Events (participants affected / at risk) | 72/476 | 79/458
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol (N=476) | Tiotropium Plus Formoterol and Placebo to QVA149 (N=458)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Amblyopia (Eye disorders) | 1 | 0
Cataract cortical (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Laryngeal fistula repair (Surgical and medical procedures) | 0 | 1
Mastectomy (Surgical and medical procedures) | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 Plus Placebo to Tiotropium and Placebo to Formoterol (N=476) | Tiotropium Plus Formoterol and Placebo to QVA149 (N=458)
Nasopharyngitis (Infections and infestations) | 42 | 53
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety